CLINICAL TRIAL: NCT02223312
Title: Phase I/II Study of Low-Dose Cyclophosphamide, Tumor Associated Peptide Antigen-Pulsed Dendritic Cell Therapy and Low Dose GM-CSF, in Patients With Progressive and/or Refractory Hematologic Malignancies
Brief Title: Therapy for Progressive and/or Refractory Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue study.
Sponsor: Kiromic BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KiroVAX002.2; BSK01 Dendritic cell vaccine (Other: Kiromic)
Record Dates: First submitted 2014-08-11; First posted 2014-08-22 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Hematologic Malignancies
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAPA-pulsed DC vaccine (Experimental): The subject will take low-dose cyclophosphamide by mouth for 5 days starting 7 days prior to the vaccine cycle. The vaccine contains 1 x 10^7 TAPA-pulsed dendritic cells and is administered SQ with low-dose GM-CSF following the low-dose cyclophosphamide cycle. A total of six (6) cycles of cyclophosphamide and six (6) DC vaccines cycles will be administered alternating every 14 days.
  Interventions: Biological: TAPA-pulsed DC vaccine

INTERVENTIONS:
Biological: TAPA-pulsed DC vaccine — A cycle of low-dose cyclophosphamide (100mg/day) by mouth for 5 days starting seven 7 days prior to the DC vaccine cycle to reduce Treg activity. Low-dose cyclophosphamide will be taken every 14 days for six 6 cycles. A total of 6 vaccines containing 1 x 10^7 TAPA-pulsed DC will be administered SQ every 14 days. The DC vaccine is given on Day 1 of the DCV cycle plus low-dose GM-CSF 50mcg/day SQ x 5 days (Day 1 to Day 4). GM-CSF is administered for 5 days to increase monocyte production and dendritic cell precursors to optimize immune responses.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Tumor Associated Peptide Antigen (TAPA) pulsed dendritic cell (DC) vaccines in the treatment of progressive and/or refractory hematologic malignancies (HM). We hypothesize that treatment of patients with relapsed and/or refractory HM, without available potentially curative treatment options, and whose neoplastic cells express at least one (1) TAPA of a defined panel of TAPAs, using low-dose cyclophosphamide (CYP) followed by an autologous, monocyte-derived, TAPA-pulsed DC vaccine and low-dose granulocyte macrophage colony stimulating factor (GM-CSF), will result in TAPA-specific T-cell responses without significant toxicities. We also hypothesize CD4+ T-cell and CD8+ T-cell responses generated against specific TAPAs may translate into clinical antitumor activity.

DETAILED DESCRIPTION:
Patients diagnosed with progressive and/or refractory hematologic malignancies, who have failed conventional therapy and have no potentially curative therapeutic options available, will be candidates for this Phase I/II study. Following confirmation of disease progression and/or refractoriness, eligible patients who agree to participate and sign a consent form will have their neoplastic cells and/or blood analyzed for the expression of a specific panel of Tumor Associated Peptide Antigens (TAPAs), including SP17, Ropporin, AKAP4, PTTG1 and Span-xb. Patients whose tumors express one (1) or more of these TAPAs will receive three (3) days of subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) to increase bone marrow production of monocytes and dendritic cell (DC) precursors, and peripheral blood mononuclear cells will be obtained by phlebotomy and/or leukapheresis for generation of autologous DCs. Patient's DCs will be generated at Kiromic's Cell Processing GMP facility, according to established Standard Operating Procedures, and activated by pulsing/loading them with the TAPA(s) relevant for each particular patient. Patients will receive five (5) days of low-dose cyclophosphamide prior to each vaccination with TAPA-pulsed DCs to decrease Treg activity. TAPA-pulsed DCs will be administered at a fixed dose of up to 1 x 107 DCs at least two (2) days following cyclophosphamide administration. DC vaccination schedule will be once every fourteen (14) days via subcutaneous (SC) and intradermal (ID) injections for a total of 6 vaccinations. Low dose GM-CSF will also be administered SC for five (5) consecutive days, starting three (3) to six (6) hours after each TAPA-pulsed DC treatment, to optimize immune response and DC viability in vivo. Patients will be followed on a weekly basis (or more frequently if required) to evaluate treatment-related toxicity. Immune responses and anti-tumor responses will be evaluated per protocol specifications. Continuation and stopping rules for the study will be defined based on toxicity/tolerability (Phase I) and/or immune efficacy (Phase II).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Patients at least eighteen (18) years of age diagnosed with the following histologically proven, progressive and/or refractory HM following standard therapy: Multiple Myeloma (MM), Hodgkins Disease (HD), Non-Hodgkins Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL), and without potentially curative therapeutic options, will be eligible.
3. Expression of one (1) or more of the following TAPAs: SP17, AKAP4, Ropporin, PTTG1 and Span-xb, by either RT-PCR and/or immunocytochemistry, Western blotting or ELISA, in neoplastic cells and/or blood.
4. Presence of measurable or evaluable disease.
5. Patients must not have any active infectious process.
6. Patients must have a negative test for HIV, Hepatitis A, B, and C.
7. Patients must not be receiving active immunosuppressive therapy.
8. Patients must have discontinued systemic antineoplastic therapy (including systemic corticosteroids) at least four (4) weeks prior to enrollment.
9. Patients may not have any known allergy to GM-CSF.
10. Patients must be willing to provide at least 250 mL, and up to 500 mL, of whole blood obtained by phlebotomy and/or consent to leukapheresis for DC generation.
11. Adequate renal and hepatic function (creatinine ≤ 2.0 mg/dl, bilirubin ≤ 2.0 mg/dl, AST and ALT ≤ 4X upper limit of normal range).
12. Adequate hematologic function (Platelets ≥ 60,000/mm3, lymphocytes ≥ 1,000/mm3, neutrophils ≥ 750/mm3, hemoglobin ≥ 10 g/dl).
13. Karnofsky performance status ≥ 70%.
14. Expected survival ≥ 6 months.
15. Patient Human Leucocyte Antigen (HLA) typing should demonstrate HLA-A*01, and/or HLA-A-*02, and/or HLA-A*24 restriction.
16. Either a female or male of reproductive capacity wishing to participate in this study must be using, or agree to use, one or more types of birth control during the entire study and for 3 months after completing the study. Birth control methods may include condoms, diaphragms, birth control pills, spermicidal gels or foams, anti-gonadotropin injections, intrauterine devices (IUD), surgical sterilization, or subcutaneous implants. Another choice is for a subject's sexual partner to use one of these birth control methods. Women of reproductive capacity will be required to undergo a urine pregnancy test before completion of the post-screening informed consent process.

Exclusion Criteria:

1. Patients without confirmed progressive and/or refractory MM, HD, NHL and CLL, or those with confirmed progressive and/or refractory MM, HD, NHL and CLL but who have a potentially curative therapeutic intervention available, are excluded from the study.
2. Patients without measurable or evaluable disease.
3. Patients receiving cytotoxic therapy, radiation therapy, immunotherapy or non-topical steroids for HM within four (4) weeks of enrollment.
4. Active immunosuppressive or cytotoxic therapy (excluding topical steroids) for any other condition.
5. Persistent fever (>24 hours) documented by repeated measurement or active, uncontrolled infection within 4 weeks of enrollment.
6. Active ischemic heart disease or history of myocardial infarction within six months.
7. Active autoimmune disease, including, but not limited to, Systemic Lupus Erythematosus (SLE), Multiple Sclerosis (MS), Ankylosing Spondylitis (AS), and Rheumatoid Arthritis (RA).
8. Pregnancy or breast feeding.
9. Active second invasive malignancy, other than basal cell carcinoma of the skin.
10. Life expectancy of less than 6 months.
11. Patients with contraindications to CYP and/or GM-CSF.
12. Patients who have received organ transplantations.
13. Patients with psychological or geographic conditions that prevent adequate follow-up or compliance with the study protocol.
14. Patients with documented primary or secondary central nervous system (CNS) involvement at any time during disease course are excluded from the study.
15. Patient with HLA-A alleles not belonging to any of the following subtypes: HLA-A*01, or HLA-A*02, or HLA-A*24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events that occur due to toxicity of low-dose CYP followed by TAPA-pulsed DC therapy and low-dose GM-CSF administration | Every 7 days

SECONDARY OUTCOMES:
Immunological efficacy as indicated by T-cell cytokine levels | up to 5 months
Immunological efficacy as determined by a positive delayed type hypersensitivity (DTH) skin test | up to 5 months
  DTH skin test will be performed 8-10 days before vaccine administration. DTH response will be evaluated again at days 28 and 70 of the trial as well as 14 and 60 days after the trial has ended.